CLINICAL TRIAL: NCT06486584
Title: Contingency Management for Problematic Behavior Reduction in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: Tulsa Day Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-005
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Bipolar Disorder; Anosognosia
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency Management (Experimental): Meet weekly for 30 minutes with their case manager to discuss progress on life goals ($10) and for having seven days with no disruptive behaviors (or "trouble-free days") per week at each visit, they will receive an additional baseline payment of $20, increasing with continued success in subsequent weeks by $1 per week.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management payment for no disruptive behaviors each week.

SUMMARY:
This study aims to determine the feasibility and effectiveness of implementing a contingency management program in a small group of mentally ill, unhoused individuals with schizophrenia or bipolar disorder and anosognosia (a lack of insight into their mental health) in the City of Tulsa. The primary objective of the study is to decrease disruptive or problematic behaviors (e.g. interactions with police, emergency services, hospitals, shelter staff, 911 calls) by unhoused individuals in the community through monetary incentives. Up to 15 participants will meet weekly for 30 minutes with their case manager to discuss progress on life goals ($10) and for having seven days with no disruptive behaviors (or "trouble-free days") per week at each visit, they will receive an additional baseline payment of $20, increasing with continued success in subsequent weeks by $1 per week.

DETAILED DESCRIPTION:
This study aims to determine the feasibility and effectiveness of implementing a contingency management program in a small group of mentally ill, unhoused individuals with schizophrenia or bipolar disorder and anosognosia (a lack of insight into their mental health) in the City of Tulsa. Tulsa's unhoused population grew nearly 7% last year to the highest numbers since the beginning of the COVID-19 pandemic according to Housing Solutions data, an organization that oversees many of the city's efforts to address homelessness. The primary objective of the study is to decrease disruptive or problematic behaviors by unhoused individuals in the community through monetary incentives.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Diagnosis of Schizophrenia Spectrum, Bipolar, or Related Disorders
3. Presence of Anosognosia (SUMD: Minimum combined score of 4 on questions 1) and 2); Recent (at least <6 months) history of disruptive behaviors (at least 1 disruptive behavior per week in >50% of weeks in the 6-month period prior to enrollment)
4. Receive case management services through TDC
5. Ability to comply with study procedures
6. Willingness to participate in contingency management intervention

Exclusion Criteria:

1. Inability to provide informed consent
2. Unstable medical conditions that would interfere with participation
3. Cognitive impairment that would interfere with participation in the study
4. History of severe aggression or violent behavior posing a risk to study staff or other participants
5. Active suicidal ideation or a history of suicide attempts within the past 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in disruptive behaviors | 6 months
  Participants will decrease the frequency of disruptive behaviors in comparison with the 6-month period immediately prior to recruitment

SECONDARY OUTCOMES:
Reduction in disruptive behaviors | 18 months
  Participants will decrease the frequency of disruptive behaviors in comparison with the 6-month period immediately prior to recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Paulus, MD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT06486584/Prot_ICF_000.pdf